CLINICAL TRIAL: NCT01012375
Title: A Phase IIa, Multi-center, Randomized, Double-blind, Placebo-controlled, Cross-Over Study to Assess the Efficacy, Safety ,Tolerability and Pharmacokinetics of Three Oral AZD1446 Dose Regimens and Placebo During 2 Weeks of Treatment in Adult Non-Users and Users of Nicotine Containing Products
Brief Title: Study to Investigate the Efficacy and Tolerability of AZD1446 in Adult ADHD Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D1950C00007
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2010-09

CONDITIONS: Adult ADHD
Keywords: Adult ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 3-(5-chloro-2-furoyl)-3,7-diazabicyclo(3.3.0)octane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): AZD1446 tid
  Interventions: Drug: AZD1446
- 2 (Experimental): AZD1446 tid
  Interventions: Drug: AZD1446
- 3 (Experimental): AZD1446 qd
  Interventions: Drug: AZD1446
- 4 (Placebo Comparator): Matching placebo capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1446 — 10 mg capsule, oral dose
  Arms: 1
Drug: AZD1446 — 80 mg capsule, oral dose
  Arms: 2
Drug: AZD1446 — 80 mg capsule, oral dose
  Arms: 3
Drug: Placebo — Matching capsule, oral dose
  Arms: 4

SUMMARY:
The purpose of this study is to determine whether 2 weeks of treatment with AZD1446 compared to placebo improves ADHD symptoms and is well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of ADHD
* Patient understands and is willing to comply with all study requirements
* Adults between the ages of 18-65 inclusive

Exclusion Criteria:

* Current psychiatric disorder other than ADHD
* Previous randomization into this study
* Women with a positive pregnancy test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
AZD1446 compared to placebo, improves ADHD core symptoms in adult non-users and users of nicotine products after 2 weeks of treatment as measured by the Conners' Adult ADHD Rating Scale-Investigator Rated (CAARS-INV) Total ADHD Symptoms score (18 item) | The CAARS-INV will be administered once at each of the following visits: Visit 1; Visit 2; Visits 3,4,5; Visit 7; Visits 8, 9, 10; Visit 12; and Visits 13, 14 and 15

SECONDARY OUTCOMES:
To evaluate the effect of AZD1446 treatment compared to placebo on ADHD symptoms as derived from the 30 item Conners' Adult ADHD Rating Scale-Investigator Rated (CAARS-INV) scoring | Visit 1; Visit 2; Visits 3,4,5; Visit 7; Visits 8, 9, 10; Visit 12; and Visits 13, 14 and 15
To assess the safety and tolerability of effects of 2 weeks treatment with AZD1446 compared to placebo. | From enrollment visit to follow up
To evaluate the pharmacokinetics (PK) of AZD1446. | Visits 2,3, 4 7, 8, 9 12, 13 and 14 PK will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Newhouse, MD, Principal Investigator — Clinical Science Research Unit, Department of Psychiatry, University of Vermont,1 South Prospect Street, Burlington, VT 05401; Bjorn Paulsson, MD, Study Director — AstraZeneca Pharmaceuticals, Kvarnbergagatan 12S-151 85, Sodertalje, Sweden
Locations (6):
- United States (6):
  - Research Site, Los Alamitos, California
  - Research Site, Fort Myers, Florida
  - Research Site, New York, New York
  - Research Site, Austin, Texas
  - Research Site, Burlington, Vermont
  - Research Site, Seattle, Washington